CLINICAL TRIAL: NCT01748487
Title: A Pilot Study of the Effect of Intravitreal Dexamethasone Implant (700 Micrograms) on Diabetic Macular Edema After Cataract Surgery
Brief Title: The Effect of Intravitreal Ozurdex on DME After Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 143BYP
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OZURDEX (Experimental): 24 patients will receive an intravitreal injection of OZURDEX at the end of cataract surgery.
  Interventions: Drug: dexamethasone intravitreal implant (OZURDEX)

INTERVENTIONS:
Drug: dexamethasone intravitreal implant (OZURDEX) — intravitreal implant
  Other Names: OZURDEX

SUMMARY:
The purpose of this study is to assess the efficacy and safety of OZURDEX (dexamethasone intravitreal implant) 0.7 mg administered immediately after phacoemulsification and intraocular lens implantation in type 1 or 2 diabetic patients to prevent the occurrence of post-surgical macular edema (ME).

Treatment group: 24 patients will receive an intravitreal injection of OZURDEX at the end of cataract surgery Patients will be seen at 1 week pre-operatively (baseline visit), and on the same day post-surgery (visit 1), at 1 week (visit 2), 1 month (visit 3) and 3 months (visit 4).

BCVA, IOP and SD-OCT will be performed at each visit.

ELIGIBILITY:
Inclusion Criteria

1. Type 1 or 2 diabetic patients for cataract surgery with > grade 3 cataract type using the Lens Opacities Classification System III. Patients with onset of diabetes before the age of 30 years and minimal or absent endogenous insulin production were classified as having type 1 diabetes. The remaining patients were classified as having type 2 diabetes.
2. Diabetics included must have at least level 20 (microaneurysms only) of diabetic retinopathy, defined by the Early Treatment Diabetic Retinopathy Study (ETDRS).
3. Patients must be healthy enough to undergo cataract surgery as decided by their physicians.
4. Patients must be 18 years older and must be able to provide informed consent.

Exclusion criteria

1. Patients with active or suspected ocular or periocular infections including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
2. Patients with advanced glaucoma.
3. Patients with known hypersensitivity to any components of this product or to other corticosteroids.
4. Patients with ACIOL (Anterior Chamber Intraocular Lens) and rupture of the posterior lens capsule
5. Patients who have aphakic eyes with rupture of the posterior lens capsule.
6. Diabetic patients without any retinopathy and those with active uncontrolled proliferative disease will be excluded. We are excluding normal retinas of diabetics since we do not feel they are at particular risk for ME when compared to those who have some form of the disease. A grading of proliferative diabetic retinopathy is based on the criteria made by the ETDRS study, which includes presence of either 1/3 optic disc neovascularization or Ã≠â√∂ optic disc area of neovascularization anywhere elsewhere in the retina.
7. Patients with clinical significant macular edema (CSME) measured with OCT prior to surgery will be excluded.
8. Panretinal photocoagulation within the prior 3 months or anticipated need for panretinal photocoagulation within the next 6 months.
9. Patients with retinal diseases, other than diabetes, that can affect ME will be excluded from the study.
10. Eyes with uveitis, a history of any other intraocular surgery or a history of uncontrolled glaucoma (baseline IOP higher than 21 mmHg or those using more than one type of glaucoma medication) or steroid responders will not be enrolled in the study.
11. Eyes with cataract precluding proper optical coherence tomography (OCT) measurement pre-operatively will also be excluded.
12. Patients who will experience longer than usual operating time, complicated surgery, rupture of the posterior capsule, and iris or corneal burns will be managed accordingly but will be excluded from the study.
13. Patients who are pregnant, breast feeding, or are unable to attend the schedules follow-up appointments will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the change from baseline for the central retinal thickness (CRT) measured by OCT at 3 months after surgery. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Brent, MD, Principal Investigator — UHN_Toronto Western Hospital
Locations (1):
- UHN, Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Calvo P, Ferreras A, Al Adel F, Dangboon W, Brent MH. EFFECT OF AN INTRAVITREAL DEXAMETHASONE IMPLANT ON DIABETIC MACULAR EDEMA AFTER CATARACT SURGERY. Retina. 2018 Mar;38(3):490-496. doi: 10.1097/IAE.0000000000001552. PMID 28196056